CLINICAL TRIAL: NCT05470218
Title: Protein, Platelet, and Monocyte
Brief Title: Leucine, MTOR and Athero
Acronym: HPL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Professor of Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HPL
Record Dates: First submitted 2022-07-13; First posted 2022-07-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Meals

STUDY DESIGN:
Intervention Model Description: Single-group crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard protein meal (Active Comparator): Participants will receive a standard protein meal, containing about 10% of energy as protein
  Interventions: Other: Meal
- High protein meal (Active Comparator): Participants will receive a high protein meal, containing about 50% of energy as protein
  Interventions: Other: Meal
- Low protein meal + leucine (Active Comparator): Participants will receive a standard protein meal, containing about 10% of energy as protein to which leucine has been added to match the total leucine content of the high protein meal
  Interventions: Other: Meal

INTERVENTIONS:
Other: Meal — Liquid mixed meal with different amounts of protein and leucine

SUMMARY:
High protein low carbohydrate diets have become popular in recent years to help facilitate weight loss. It is controversial if these diets are associated with an increased risk of cardiovascular disease. Recent work in mice has implicated monocytes/macrophages and mTOR signaling as the culprit cell type driving the increased cardiovascular risk with high protein diets. We aim to build on this preclinical research by evaluating the effects of liquid meals with different protein and leucine (a potent mTOR activator) contents on circulating human monocytes and platelets. Study participants will be given either a low protein liquid meal, a high protein liquid meal, or a low protein liquid meal with additional leucine. Blood will be collected from study participants just just prior to and for several hours after ingestion of the meals. Activation of amino acid-dependent signaling pathways (particularly mTOR) and downstream sequelae will be evaluated in the isolated monocytes and platelets.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able to drink milk-based liquid mixed meal

Exclusion Criteria:

* Current Pregnancy
* Allergies to meal ingredients
* History of Diabetes
* History of Heart Disease
* History of High blood pressure
* History of Stroke
* History of Cancer
* History of Organ transplant
* Taking Rapamycin/Sirolimus
* Taking Torisel/Temsirolimus
* Taking Afinitor/Everolimus
* Taking any statin medication

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
p-mTOR in monocytes | change from before meal at 1 hour and 3 hours, compared to before

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request beginning 12 months and ending 36 months following article publication
Supporting Information: Study Protocol
Time Frame: beginning 12 months and ending 36 months following article publication